CLINICAL TRIAL: NCT00872040
Title: Observational Study on the Effect of Delivery Mode on Inter Personal Relationship, Sexual Function and Pelvic Floor Activity
Brief Title: The Effect of Delivery Mode on Inter - Couple Relationship, Sexual Function and Pelvic Floor Activity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Menachem Alcalay, Head - Urogynecology Service, Chaim Sheba Medical Center
Other Study IDs: SHEBA-09-5177-MA-CTIL
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Pregnancy
Keywords: Sexual function; Pelvic floor disorders; Delivery mode
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nuliparous women and their husbands: Women in their first pregnancy with their husbands
  Interventions: Other: Ultrasound assessment of pelvic floor

INTERVENTIONS:
Other: Ultrasound assessment of pelvic floor — Sample of women will undergo ultrasound examination of their pelvic floor before and after delivery. The assessment will be performed by transperineal probe.
  Other Names: Ultrasound examination of pelvic floor

SUMMARY:
Pregnancy and delivery have a major impact on couple's inter personal relationship. Different modes of delivery have different effect on pelvic floor function, and it is known that instrumental vaginal deliveries have the worse effect, though various common anatomical injuries have been described following vaginal delivery. Pelvic floor dysfunction has the potential to ameliorate sexual function, and the investigators hypothesis is that the impact of delivery on pelvic floor disorders following delivery will have a direct effect on sexual malfunction and interpersonal relationship. The purpose of this study is to evaluate the effect of delivery mode of primiparous women on inter couple relationship , their sexual function and the female pelvic floor activity. The couples will be followed from the second trimester of the pregnancy by validated specific questionnaires, assessing the couple's satisfaction of their marriage, intimacy in their relationship, their sexual behavior and pelvic floor function. After delivery, the parameters of the parturition will be recorded, and the couples will be interviewed 6 months following delivery. Apart from questionnaires, sample of the participated women will be assessed by ultrasound examination of the pelvic floor.

DETAILED DESCRIPTION:
Pregnant women in their first pregnancy and their husbands will be recruited from 14th week of gestation. The couples will be followed by validated specific questionnaires, such as Couple Satisfaction Index (CSI), Isreali Sexual Behavior Inventory (ISBI), Pelvic Floor Distress Inventory (PFDI)and Pelvic Floor Impact Questionnaire (PFIQ) assessing the couple's satisfaction of their marriage, intimacy in their relationship, their sexual behavior and pelvic floor function. After delivery, the parameters of the parturition will be recorded, and the couples will be interviewed 6 months following delivery. Apart from questionnaires, sample of the participated women will be assessed by ultrasound examination of the pelvic floor, demonstrating the continuity of pelvic floor muscles and their function.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in their 1st pregnancy
* Married couples in their 1st marriage

Exclusion Criteria:

* Chronic GIT disease
* Endometriosis
* Chronic GUT disease
* Psychiatric disease
* Known sexual dysfunction

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who attend primary care antenatal clinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-10 (Estimated); Study Completion 2011-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Oria Tishbi, PhD, Study Chair — School of Social Work, Hebrew University, Jerusalem
Locations (1):
- Antenatal primary care clinic, Kfar Saba, Israel